CLINICAL TRIAL: NCT06798493
Title: Validation of the CRPS Severity Score-Self Report
Brief Title: CSS-SR Validation Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1529
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Complex Regional Pain Syndrome; Pain
Keywords: CRPS; Complex Regional Pain Syndrome; self-report; Complex Regional Pain Syndrome Severity Score (CSS)
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CRPS group: Patients suspected or diagnosed with unilateral CRPS type I or II of the upper or lower extremity
  Interventions: Other: Complex Regional Pain Syndrome (CRPS) Severity Score - Self Report
- Non-CRPS group: Patients suspected or diagnosed with non-CRPS-related pain of the upper or lower extremities
  Interventions: Other: Complex Regional Pain Syndrome (CRPS) Severity Score - Self Report

INTERVENTIONS:
Other: Complex Regional Pain Syndrome (CRPS) Severity Score - Self Report — Self-report tool in a questionnaire format to capture CPRS Severity Score.

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is an orphan condition with no interventions proven effective in large-scale clinical trials. In-person clinical evaluations are required to make a CRPS diagnosis and determine study eligibility, making recruitment for CRPS trials challenging. To address this barrier, we will validate a self-report measure of CRPS symptom severity suitable for remote administration that was created by colleagues at Vanderbilt University.

The aim of this study is to evaluate the correspondence at the item and total score level between the proposed self-report measure (CRPS Severity Score-Self Report; CSS-SR) and an existing validated measure of CRPS signs and symptoms derived from clinical history and physical examination data (CSS-Clinician version) and evaluate its diagnostic accuracy relative to clinically determined, criterion-based CRPS diagnosis using the Budapest criteria.

DETAILED DESCRIPTION:
Complex Regional Pain Syndrome (CRPS) is a chronic pain condition characterized by spontaneous pain, allodynia and hyperalgesia, edema, vasomotor and sudomotor changes, and motor and trophic changes. It usually begins regionally in a single limb after injury or surgery, and inflammatory, autonomic, and central mechanisms all appear to contribute to differing degrees. There are currently no treatments for CRPS proven effective in large scale clinical trials.

CRPS is considered an orphan condition by the U.S. Food and Drug Administration, and as such, acquiring adequate sample sizes for definitive clinical trials is challenging. One barrier to recruitment into CRPS research studies is the need to conduct in-person evaluations to screen for presence of current CRPS clinical features and determine CRPS diagnostic status. Unlike conditions such as chronic low back pain, which can be identified with high accuracy based on questions that can be administered remotely (i.e., pain intensity, location, frequency, and impact), diagnosing CRPS using the 2012 International Association for the Study of Pain (IASP) criteria (i.e., the Budapest criteria) requires that a history and physical examination be conducted. This situation is similar to that formerly encountered in fibromyalgia studies prior to publication of the modified American College of Rheumatology 2010 criteria (i.e., diagnosis was based on clinical tender point evaluation), a barrier ultimately overcome by publication of the validated 2010 self-report diagnostic screening criteria that could be administered remotely.

Our collaborators developed a self-report measure suitable for remote delivery to assess CRPS-related symptoms. They evaluated the diagnostic accuracy of a self-report version of the CRPS Severity Score (CSS-SR) and assessed its validity relative to the original CSS based on clinician evaluation (CSS-Clinician) in 112 patients undergoing total knee arthroplasty (TKA). In this study we will recruit patients with pain in an extremity at the outpatient chronic pain clinic at 75th street and will ask patients to complete the CSS-SR while the clinician evaluates the participant against the Budapest CRPS diagnosis criteria per usual care. Data (no identifiers) will be shared with our collaborator who will analyze and combine the findings from his TKA cohort with our outpatient chronic pain cohort to understand the external validity of the CSS-SR.

The proposed content of the self-report version of the CSS (CSS-SR) was rationally developed by creating lay language items designed to parallel the diagnostic symptoms assessed in the standardized clinician-obtained history that provides the basis for the symptom component of the CSS-Clinician. Thirteen questions in yes/no (presence/absence) checklist format assess presence of symptoms in the following areas: more prolonged or severe pain than expected, allodynia/hyperalgesia, skin temperature changes, skin color changes, edema, sweating changes, trophic changes (skin, hair, nails), tremor, dystonia, weakness, and range of motion limitations.

Scoring of the CSS-SR parallels scoring of the CSS-Clinician, with items coded as 1 for "Yes" and 0 for "No", with responses summed to create a total CSS-SR score potentially ranging from 0-13.

For the current validation study, CSS-SR items referred specifically to the "affected limb" to ensure that participants describe symptoms in the same body region as reflected in the assessment used to derive the CSS-Clinician.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Suspected or diagnosed with unilateral CRPS type I or II of the upper or lower extremity
* Suspected or diagnosed with non-CRPS-related pain of the upper or lower extremities

Exclusion Criteria:

* Bilateral CRPS
* Total knee arthroplasty as the inciting event of CRPS
* Less than 18 years of age
* Non-English speaking
* Inability to comprehend study protocol and questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital for Special Surgery Outpatient Pain Management Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Concordance between CSS-Clinician and CSS-SR total scores | Date of enrollment
  Concordance between CSS-Clinician total scores, which will be on a numerical scale potentially ranging from 0-16, and CSS-SR total scores, which will be on a numerical scale potentially ranging from 0-13. Higher scores indicate greater CRPS symptom severity while lower scores indicate a lesser degree of symptom severity. Concordance (corrected for chance agreement) between CSS-Clinician and CSS-SR items and total scores will be assessed using intraclass correlations (ICCs; two-way random effects model; potential range = -1.00 to 1.00). Strength of agreement will be evaluated for descriptive purposes based on published recommendations: < 0.50 = poor agreement, 0.50 - 0.75 = moderate agreement, 0.76 - 0.90 = good agreement, and >0.90 = excellent agreement. All analyses will use the maximum number of cases available with a two-sided p<0.05 criterion for statistical significance.

SECONDARY OUTCOMES:
Diagnostic accuracy relative to clinically-determined, criterion-based CRPS diagnosis using the Budapest criteria | Date of enrollment
  Rates of CRPS diagnoses on both the CSS-Clinician and CSS-SR will be summarized as frequencies of positive and negative diagnoses.
  Cut scores on the CSS-SR for use in determining its accuracy as a screening tool for predicting dichotomous criterion-based CRPS diagnosis will be generated by inspection of receiver operating characteristic (ROC) curves and associated sensitivity/specificity values. All analyses will use the maximum number of cases available with a two-sided p<0.05 criterion for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sideris, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan will be finalized with our collaborators at study completion.

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Bruehl S. An update on the pathophysiology of complex regional pain syndrome. Anesthesiology. 2010 Sep;113(3):713-25. doi: 10.1097/ALN.0b013e3181e3db38. PMID 20693883